CLINICAL TRIAL: NCT03894397
Title: Evaluating Unilateral Deep Brain Stimulation (DBS) of the Bed Nucleus of the Stria Terminalis (BNST) in Patients With Obsessive Compulsive Disorder (OCD)
Brief Title: Evaluating Unilateral Deep Brain Stimulation in Patients With Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kelly Luyck, PhD, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: S62175
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: (Unilateral) Deep brain stimulation; Anxiety; Mood
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: We will evaluate the effect of unilateral and bilateral stimulation of the BNST. Four conditions will be evaluated: left BNST stimulation, right BNST stimulation, bilateral BNST stimulation or no stimulation (OFF). Note that the order of these conditions is stratified beforehand (www.random.org). Each condition takes around 15 minutes.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both the patient and the psychiatrist are blinded during the cross-over phase, until the end of the study. The investigator who will evaluate behavior from the videorecordings, will also be blinded.
  Unblinded are: the principal investigator (who has access to all data) and the technical staff in charge of stimulation settings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Stimulation of left BNST (Experimental)
  Interventions: Device: Electrical stimulation of the BNST
- Stimulation of right BNST (Experimental)
  Interventions: Device: Electrical stimulation of the BNST
- Stimulation of bilateral BNST (Experimental)
  Interventions: Device: Electrical stimulation of the BNST
- Stimulation OFF (Placebo Comparator)
  Interventions: Device: Electrical stimulation of the BNST

INTERVENTIONS:
Device: Electrical stimulation of the BNST — Electrical stimulation of the BNST

SUMMARY:
The investigators previously showed that deep brain stimulation (DBS) in the bed nucleus of the stria terminalis (BNST) reduces symptoms in patients with severe obsessive-compulsive disorder (OCD). Although most patients now receive bilateral stimulation, multiple studies suggest that stimulation of the left BNST might be equally effective.

In this study, the investigators will evaluate the effect of unilateral stimulation in OCD patients who currently receive bilateral BNST stimulation to treat their symptoms. We hypothesize that unilateral stimulation of the left BNST will reduce anxious and depressive symptoms, compared to no stimulation.

The study entails a double-blinded, randomized cross-over design during which every patient undergoes four stimulation conditions: stimulation of the left, right or bilateral BNST, or no stimulation. During every condition, which takes about fifteen minutes, the patient is exposed to an individually determined stimulus that normally elicits OCD-related symptoms. The patients are then asked to fill out a short questionnaire to evaluate the severity of their symptoms during the four conditions. At the end of the cross-over phase, the stimulation parameters of each patient are restored.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of obsessive-compulsive disorder
* Implanted with DBS system in the bilateral BST (or max. 4mm removed from the BST outline)
* At least three months of chronic BST stimulation
* Compulsive behavior can be provoked within a clinical setting

Exclusion criteria:

* Personality changes evoked by chronic DBS
* Cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) ratings of mood and anxiety/stress | After 15 minutes of stimulation
  For every question on the VAS, there will be a line of 10 centimeters as an outcome measure. The patient will place a mark on this line, in correspondence to their symptoms. The minimum is 0%, which corresponds to no symptoms at all. The maximum is 100% (marker at the end of the 10 centimeter line), and indicates the most severe symptoms. Every millimiter that the mark is removed from the left boundary of the line, is considered as 1%. Measurements of mood and anxiety/stress will be scored using 2 VAS scales. We will only look at sub score, not total scores. A higher score corresponds to more severe symptoms. By using a continuous line as an outcome rather than fixed numbers (1-2-3-...), our rating is far more sensitive to small deviations in how symptoms are experienced.

SECONDARY OUTCOMES:
VAS ratings of obsessive thoughts, urge to perform compulsive behavior, avoidance and global wellbeing | After 15 minutes of stimulation
  For every question on the VAS, there will be a line of 10 centimeters as an outcome measure. The patient will place a mark on this line, in correspondence to their symptoms. The minimum is 0%, which corresponds to no symptoms at all. The maximum is 100% (marker at the end of the 10 centimeter line), and indicates the most severe symptoms. For global wellbeing, a higher score corresponds to better therapeutic effects. Every millimiter that the mark is removed from the left boundary of the line, is considered as 1%. Obsessive thoughts, urge to perform compulsions, avoidance and global wellbeing will be measured using four separate VAS scales. We will only look at sub score, not total scores. By using a continuous line as an outcome rather than fixed numbers (1-2-3-...), our rating is far more sensitive to small deviations in how symptoms are experienced. For obsessive thoughts, urge to perform compulsions and avoidance, a higher score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University Leuven, Leuven, Vlaams-Brabant, Belgium